CLINICAL TRIAL: NCT04506177
Title: E-PACT: Extension Trial of Permanent Versus Delayed-absorbable Monofilament Suture for Vaginal Graft Attachment During Minimally-invasive Total Hysterectomy and Sacrocolpopexy
Brief Title: Permanent Versus Delayed-Absorbable Monofilament Suture
Acronym: E-PACT
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00036663
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Hysterectomy; Sacrocolpopexy
Keywords: Pelvic Organ Prolapse; Vaginal mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Permanent Sutures: Women who previously received (in the PACT Study Trial) minimally-invasive total hysterectomy and sacrocolpopexy (SCP) with a light-weight polypropylene mesh (Upsylon™ y-mesh) using permanent (polytetrafluoroethylene, Gore-Tex) suture for vaginal mesh attachment
- Delayed Absorbable Monofilament Sutures: Women who previously received (in the PACT Study Trial) minimally-invasive total hysterectomy and sacrocolpopexy (SCP) with a light-weight polypropylene mesh (Upsylon™ y-mesh) using delayed absorbable monofilament (polydioxanone, PDS) suture for vaginal mesh attachment

SUMMARY:
This is an extension study of a prospective, multicenter, randomized, single-blind trial whose purpose is to compare mesh-related complications and effectiveness of pelvic organ prolapse (POP) repair in women undergoing minimally-invasive total hysterectomy and sacrocolpopexy (SCP) with a light-weight polypropylene mesh (Upsylon™ y-mesh) using permanent (polytetrafluoroethylene, Gore-Tex) versus delayed absorbable monofilament (polydioxanone, PDS) suture for vaginal mesh attachment through at least 3 years after surgery.

DETAILED DESCRIPTION:
This is an extension study of a randomized controlled trial that will be conducted at the same 5 clinical sites as the primary study - All subjects who participated in the original randomization and did not withdraw from the study are eligible for the extension study including those with a history of secondary treatment following PACT RCT study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have participated in the PACT Study Trial (Permanent Versus Delayed-absorbable Monofilament Suture for Vaginal Graft Attachment During Minimally-invasive Total Hysterectomy and Sacrocolpopexy: A Randomized Clinical Trial)

Exclusion Criteria:

* Patient is not willing to sign consent
* Patient does not want to fill-out questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with the history of hysterectomy and sacrocolpopexy
Study Population: Study Patients who have participated in the PACT Study Trial at one of the following Research Sites:
  1. Wake Forest University, Winston-Salem (22 subject participants)
  2. University of North Carolina, Chapel Hill
  3. Northwestern Medical Center, Chicago
  4. Augusta University, Augusta
  5. Atrium Health, Charlotte
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Vaginal Mesh or Suture Exposure | Post Procedure Evaluation at Minimum 2 years
  Total number of participants (96% with permanent and 86% absorbable suture) will be examined and evaluated for vaginal mesh and/or suture exposure at 2 years or grater time period. Exposure of the suture or mesh will be defined upon the visual examination in the clinic, It is expected to identify <10% patient population during examination
Vaginal Mesh or Suture Exposure | Post Procedure Evaluation at 3 years
  Total number of participants (96% with permanent and 86% absorbable suture) will be examined and evaluated for vaginal mesh and/or suture exposure at 3 years or grater time period. Exposure of the suture or mesh will be defined upon the visual examination in the clinic, It is expected to identify <10% patient population during examination

SECONDARY OUTCOMES:
Anatomic success | Post Procedure Evaluation at Minimum 2 years and 3 years
  Leading edge of the prolapse is at or above the hymen to be evaluate among expected 200 participants. POP-Q assessment will be performed with surgical success being defined as apical descent less than 50% of total vaginal length
Subjective success | Post Procedure Evaluation at Minimum 2 years and 3 years
  PFDI-20 (Pelvic Floor Disability Index) - Patient denies symptoms of vaginal bulging per question 3, answering "No" or "Yes". Response "Yes" leads to 4 probabilities of bothersome of condition from none to quite a bit (3 scales of symptoms and 0 as "Not at all"). Higher the value indicates a greater degree of bother. It is expected to have <10% to have bulge symptoms by the end of the study.
Assessment for re-intervention or re-surgery for recurrence of persistence of POP | Post Procedure Evaluation at Minimum 2 years and 3 years
  No necessary use or additional surgical treatment for prolapse at any time after the initial procedure among expected 200 participants who have had participated in the original PACT study trial. Usage of pessary will be accounted as retreatment with expected <1% patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Matthews, MD, Principal Investigator — Wake Forest Health Sciences
Locations (5):
- United States (5):
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No